CLINICAL TRIAL: NCT02172807
Title: A Multiple Dose Comparison of 18 µg, 36 µg of Ba679BR (Tiotropium) Inhalation Capsules and Oxitropium Metered Dose Inhaler (2 Puffs of 100µg) in a 4-week, Double-Blind, Double-Dummy, Safety and Efficacy Study in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety of Ba679BR Powder Inhalation in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.226
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — oxitropium

ARMS (3):
- Tiotropium low & Placebo (Experimental): Tiotropium 18 µg inhalation capsule and Placebo MDI
  Interventions: Drug: Tiotropium low; Drug: Placebo MDI
- Tiotropium high & Placebo (Experimental): Tiotropium 36 µg inhalation capsule and Placebo MDI
  Interventions: Drug: Tiotropium high; Drug: Placebo MDI
- Oxitropium & Placebo (Active Comparator): Oxitropium MDI (100 µg/puff) and Placebo inhalation capsules
  Interventions: Drug: Placebo inhalation capsule; Drug: Oxitropium

INTERVENTIONS:
Drug: Tiotropium low — Tiotropium 18 µg inhalation capsule
  Arms: Tiotropium low & Placebo
Drug: Tiotropium high — Tiotropium 36 µg inhalation capsule
  Arms: Tiotropium high & Placebo
Drug: Placebo MDI — Placebo metered dose inhaler (MDI)
  Arms: Tiotropium high & Placebo; Tiotropium low & Placebo
Drug: Placebo inhalation capsule
  Arms: Oxitropium & Placebo
Drug: Oxitropium — Oxitropium MDI (100 µg/puff)
  Other Names: Tersigan®
  Arms: Oxitropium & Placebo

SUMMARY:
Study to investigate the efficacy and safety of Ba679BR powder inhalation during the continuous once/day administration to the patients with COPD using oxitropium bromide (Tersigan® aerosol) as the comparator drug.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of COPD (chronic bronchitis, and emphysema) with stable symptoms:

* Screening FEV1.0 ≤70% of predicted normal vale and screening FEV1.0/FVC ≤70% (the baseline FEV1.0 should also be ≤70% of predicted normal value on the initial day of administration)
* Smoking history ≥ 10 pack-years (a peak-year is 20 cigarettes per day for one year or equivalent)
* Male or female patients 40 years of age or older

Exclusion Criteria:

* History of bronchial asthma
* History of an atopic disease such as allergic rhinitis
* Total blood eosinophil count ≥ 600/µL
* Patient treated with antiallergic drugs or anti-histamine drugs
* Patients using oral corticosteroid medication at unstable doses (i.e. less than one month on a stable dose) or at a dose in excess of the equivalent of 10 mg of prednisolone per day
* Patients using inhaled steroid, oral β2 stimulant, theophylline preparation, expectorant or macrolide antibiotic at unstable doses (i.e. less than one month on a stable dose)
* Patients using an ACE inhibitor at unstable doses (i.e. less than one month on a stable dose)
* Patients with known narrow-angle glaucoma
* Patients with known symptomatic prostatic hypertrophy
* Patients with known hypersensitivity to anticholinergic drugs, lactose or any other components of the inhalation capsule delivery system
* Patients with significant diseases who in the opinion of the investigator were not eligible for the study
* Patients with clinically significant abnormal baseline laboratory test values (hematology, blood chemistry, urinalysis). Patients with serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamic-pyruvic transaminase (SGPT) twice the upper limit of the normal range, bilirubin 150% or creatinine 125% of the upper limit of the normal range were excluded
* Patients with a recent history (i.e. within the 3 months prior to the screening visit) of myocardial infarction or heart failure
* Patients with any cardiac arrhythmia requiring drug therapy
* Patients who were treated with Patients who were treated with β-blockers-blockers
* Patients with regular use of daytime oxygen therapy
* Patients with known active tuberculosis or with obvious sequela of tuberculosis
* Patients with a history of cancer within the last 5 years. Patients with treated basal cell carcinoma were allowed
* Patients with a history of cystic fibrosis or bronchiectasis
* Patients with upper respiratory tract infection in the past one month prior to the screening visit or during the baseline period
* Patients who had taken an investigational drug within one month or six half lives (whichever is greater) prior to the screening visit
* Pregnant or nursing women or women of childbearing potential
* Other than the above, patients who in the opinion of the investigator were not eligible for the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2000-12; Primary Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Trough forced expiratory volume in one second (FEV1.0) response | Day 1, week 2 and 4

SECONDARY OUTCOMES:
FEV1.0 response at 1 hour after administration | Day 1, week 2 and 4
Trough forced vital capacity (FVC) response | Day 1, week 2 and 4
FVC response at 1 hour after administration | Day 1, week 2 and 4
Peak expiratory flow rate (PEF) | in the morning and at evening every day until week 4
COPD symptom scores | until week 4
Frequency of rescue use of β2 stimulant | until week 4
Patient's impression | week 4
Physician's global evaluation | week 4
Occurrence of Adverse Events | up to 4 weeks
Change from baseline in blood pressure | Baseline, week 4
Change from baseline in heart rate | Baseline, week 4
Changes in ECG findings | Baseline, week 4
Changes from baseline in laboratory values | Baseline, week 4